CLINICAL TRIAL: NCT04287751
Title: PROXIMO: A Cohort Study to Investigate the Incidence of Obstructive Sleep Apnoea Using Prolonged Overnight Oximetry in an Unselected Population Referred to Secondary Care Reporting Excessive Daytime Sleepiness
Brief Title: Prolonged Overnight Oximetry in Obstructive Sleep Apnoea
Acronym: PROXIMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Somerset NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Justin Pepperell, Consultant Physician in Respiratory and General Medicine; Honorary Senior Lecturer University of Exeter; Director of Department of Clinical Research; Secretary of the British Thoracic Society, Somerset NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/LO/0055
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnoea; Overnight Oximetry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Recruiting participants undergoing overnight oximetry on a single night to have additional 4 nights of recording with a prolonged recording oximeter device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overnight Oximetry (Other): Participants record simultaneously overnight oximetry on night 1 and continue with prolonged recordings alone for a total of 4 nights
  Interventions: Device: CheckMeO2 Oximeter

INTERVENTIONS:
Device: CheckMeO2 Oximeter — Simultaneous recording with a current standard oximeter (Minolta i300) and prolonged recording device. Comparison of data from first night and incidence of obstructive sleep apnoea identified from additional nights of recording identified.

SUMMARY:
This study is looking at the way in which patients with obstructive sleep apnoea (OSA) are diagnosed. The investigators current practice is to offer patients who are referred to the sleep centre with possible sleep apnoea a single night's oximetry recording. A decision is then made based on this screening test as to whether the patient has OSA, does not have OSA or requires a further investigation. There can be significant variation in the severity of OSA between nights. This study is designed to investigate if recording data from multiple nights will give any better indication on the presence and severity of obstructive sleep apnoea. Patients referred for overnight oximetry recordings that report excessive daytime sleepiness are eligible to enter the trial.

On enrolment participants will all undergo a single night recording with the oximetry device currently in use by the recruiting sleep centre. In addition they will be asked to wear the prolonged recording oximeter (PRO) that allows for multiple nights data to be stored, and continue wearing this for a total of four nights. On returning both oximetry devices, this data will then be analysed and if it demonstrates evidence of OSA participants will return to the standard clinical pathway and be offered a trial of treatment with continuous positive airway pressure (CPAP) therapy.

If no evidence of OSA is seen participants will also revert back to the standard clinical pathway, which may involve a further inpatient sleep investigation being arranged.

The number of patients identified as having OSA based on the single first night recording will be compared to those identified as having OSA only after the additional nights recording.

All participants will return to the current standard pathway of care on leaving the trial.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a common condition, effecting an estimated 1.5 million people in the UK and it is believed up to 80% of them may be undiagnosed [1]. During sleep the muscles supporting the upper airway tend to relax and the throat narrows. In patients with OSA the narrowing leads to collapse and pauses in breathing. These pauses in breathing are accompanied by a decrease in arterial oxygen saturation and to overcome the airway collapse the body responds by producing a surge in the sympathetic nervous system. This has the effect of stimulating the pharyngeal muscles to reopen the throat but also causes an increase in heart rate, blood pressure and disrupts the sleep cycle waking the patient up. These repeated disruptions to sleep leads to the patient feeling unrefreshed by sleep, excessively sleepy during the day and at increased risk of a sleepiness-related accident. The repetitive surges in the sympathetic nervous system also contributes to the risk of long term cardiovascular disease. The frequency with which these events occur determines the severity of obstructive sleep apnoea, less than 5 events per hour is considered normal, 5-15 mild, 15-30 moderate and more than 30 severe disease. However the disease severity does not correlate with the degree of symptoms [2] meaning it is important to identify patients even if they have mild and moderate disease.

OSA is effectively treated with continuous positive airway pressure (CPAP) therapy. These machines blow air into the throat through a nose or face mask. This helps to splint the airway open and reduce the disruption to sleep. CPAP is an effective therapy improving sleepiness, snoring, mood and reduces the long term risk of cardiovascular disease seen in untreated patients with OSA.

Full inpatient polysomnography testing is the gold standard investigation for diagnosis and exclusion of OSA [3]. However because polysomnography generally requires a hospital bed, significant technical input to set up and is time intensive to report it is impractical for the large numbers of patients referred to sleep services to undergo this test. Overnight oximetry recording has been established as an effective alternative for screening patients and identifying OSA in many sleep centres [4-6].

For a single test to be effective it needs to be highly sensitive and the condition being investigated should be stable. However significant variation in the severity of obstructive sleep apnoea has been demonstrated from night to night in individual patients [7, 8]. Therefore using oximetry or even polysomnography recording for a single night may not truly reflect the overall condition. Patients with mild and moderate disease show the most significant variations on a night to night basis, as the oxygen desaturation index (ODI, number of times the oxygen saturations dip per hour) rises, i.e. more severe OSA, less night to night variability is observed [9]. When patients with previously diagnosed OSA are withdrawn from CPAP treatment and overnight oximetry performed for two weeks only 22% of participants consistently remain within one severity category. The majority of these patients were in the severe category. Other studies have shown 40-50% of patients changing severity category in two to four nights recordings [7, 10] and that 16-20% of patients would not have received CPAP treatment based on a single night study but did so after repeating between one to three studies [10, 11].

The most clinically relevant distinction to make is between no OSA and mild and moderate OSA as this determines whether a trial of CPAP therapy would be offered. These previous trials suggest it is within this milder spectrum of the disease where a single night's oximetry recording is least reliable and more than one night's recording may be required.

Despite CPAP being a very successful treatment for OSA, adherence rates to treatment are variable [12, 13]. It has also be shown that adherence correlates with OSA severity [14]. In part this poor adherence to treatment suggests imperfect identification of patients. The investigators hypothesise that the current oximetry screening of a single night may not be effectively identifying all those patients who may benefit from CPAP. The investigators aim to identify how many additional patients are identified as having OSA with prolonged, multi-night recordings. A longer period of oximetry recording may improve the identification of those patients who may benefit from CPAP and may help to identify factors that predict a poorer response to CPAP therapy. Therefore this study will follow-up patients to see if those identified by prolonged oximetry screening tests leads to improved adherence to CPAP.

Two different oximeters are used in this study. The Minolta i300 was chosen as it is the current device used within the investigators clinical service. This is not being used for prolonged recordings as the battery life makes it impractical to be used for more than two nights recording. Therefore the CheckMeO2 oximeter was chosen; this has a rechargeable battery and sufficient memory capacity to be used for the required 4 nights of recording.

The CheckMe O2 device records oxygen saturations to nearest whole number every 4 seconds versus the Minolta device recording to one decimal place every second. It is felt that as the average length of a desaturation in obstructive sleep apnoea is 15-20 seconds the CheckMe O2 device should be sufficiently accurate to detect OSA but by performing a simultaneous recording during the first night the investigators hope to establish if this frequency of recording is sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and give informed consent to participate
* Male or Female aged 18 years or older
* Referral letter or request to sleep service reports an Epworth Sleepiness Score of greater than 9 or reason for the referral is 'excessive daytime sleepiness'

Exclusion Criteria:

* Significant cardiovascular or respiratory co-morbidities
* Suspected hypoventilation or sleep disordered breathing
* Previously used Non-invasive ventilation
* In the Investigators opinion an alternative diagnostic test should be offered as first line e.g. referral information suggests an inpatient sleep study is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of OSA on 1 night vs 4 nights Oximetry | 4 days
  To compare the incidence of OSA using current single night recording versus multiple night recordings

SECONDARY OUTCOMES:
To compare the adherence rates to CPAP at 1 month follow-up | 1 month
  Compare the adherence rates to CPAP between those identified after 1 night compared to those identified after a prolonged recording. Adherence will be measured using CPAP machine usage records accessed at the one month follow-up. The mean hours used per night will be compared between the two groups
To assess the tolerability of prolonged oximetry screening for patients | 4 days
  Patient questionnaire feedback comparing tolerability of prolonged recordings. A 10cm Visual analogue scale will be used to assess how tolerable and easy to use each oximeter device is. Higher scores suggest the device is more tolerable.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Pepperell, Principal Investigator — Somerset NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No